CLINICAL TRIAL: NCT04255160
Title: Impact of Estradiol on Endothelial Function in Peri-Menopausal Women
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Megan M. Wenner, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1508142; R01HL146558 (NIH)
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Perimenopause; Vasodilation; Estrogen
Keywords: Perimenopause; Vasodilation; Estrogen
MeSH Terms: conditions — Aneurysm | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Estradiol (Experimental): Transdermal estradiol (0.1mg/day patch)
  Interventions: Drug: Estradiol (mylan or vivelle dot patch)
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Estradiol (mylan or vivelle dot patch) — Transdermal estradiol (0.1mg/day patch) will be used by women for 7 days. Administration of the patch will follow the package guidelines to change the patch after 3-4 days of use.
  Arms: Estradiol
Other: Placebo — A placebo patch that is visually similar to the estradiol patch will be used for the group not receiving estradiol.
  Arms: Placebo

SUMMARY:
The purpose of this study is to identify the impact of estradiol (E2) on the mechanisms that regulate vascular endothelial function in peri-menopausal (PERI) women. This study is the first step in understanding factors contributing to endothelial dysfunction in women with advancing reproductive age and in response to E2 administration.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in women. Although overall CVD-related mortality has declined, there has been an increase in CVD mortality in women aged 35-54 years, prior to menopause. It is unclear what contributes to this increased mortality rate, and is a significant problem for women's health. Endothelial function is considered a biomarker of cardiovascular health; declines in endothelial function are considered a precursor to the development of atherosclerosis and CVD. Thus, changes in endothelial function in women as they advance through reproductive stages towards menopause may play a role in the greater prevalence of CVD mortality. However, very few studies have focused on cardiovascular health in women leading up to menopause, during the PERI transition. The PERI period is a critical time point where reproductive hormones and ovarian function change rapidly. Recent data demonstrate that endothelial function begins to decline during PERI. Furthermore, despite women being of similar biological age, significant differences in endothelial function were noted when classified based on reproductive age - specifically between early PERI and late PERI. These data show that the decline initially occurs in the early PERI phase, making this a key time point for intervention to offset the future development of CVD. Our central hypothesis is that increased Endothelin-1 (ET-1) and a loss of Endothelin-1 B (ETB) mediated vasodilation play a primary role in contributing to impaired endothelial function with advancing reproductive age. We will assess macro- and micro- vascular endothelial function, assess intracellular ET-1 protein and ETB receptor expression in harvested endothelial cells from peripheral veins, and use the cutaneous circulation as an in vivo model to explore the receptor mechanisms (ETBR and ETAR) in early and late PERI in response to E2 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Peri-menopausal women between 40-58 years of age with variable cycles as defined by increase in cycle length of greater than 7 days within ten consecutive cycles, or amenorrhea for more than 2 months, but less than 12 months.

Exclusion Criteria:

* Women who are pregnant, planning on becoming pregnant, or are breast feeding;
* Women who have a history of cardiovascular disease, blood clots (e.g, pulmonary embolism or deep vein thrombosis), stroke, cancer, or liver disease;
* Women who have a body mass index less than 18 or greater than 35kg/m2;
* Women who use tobacco products;
* Women who's blood pressure is greater than 140/90 mmHg, have been diagnosed by a physician with hypertension or are taking medication for high blood pressure;
* Women who have a neurological disease, or diabetes;
* Women who have had a hysterectomy or have used hormones (birth control or hormone replacement) within the past 3 months;
* Women who have a latex allergy.

Ages: 40 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Vascular Endothelial Function (Flow mediated dilation or FMD) | Change in FMD from Baseline to Day 7
  The capacity of the large and small blood vessels to dilate.

SECONDARY OUTCOMES:
Endothelial Cell Protein Expression | Change in fluorescent intensity from Baseline to Day 7
  Venous endothelial cells will be harvested from peripheral veins of women during the hormone intervention and stained for expression of ET-1 and ETB receptors.
Endothelin Receptor Responses | Change from Baseline to Day 7
  The contribution of Endothelin A (ETA) and Endothelin B (ETB) receptors on changes in endothelial function will be assessed in the cutaneous circulation via microdialysis. Blood flow responses to local heating will be assessed under control and blockade sites in women during estradiol or placebo administration.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No